CLINICAL TRIAL: NCT04655885
Title: Effect of an Individualized Protocol Based on Cardiac Output Optimization Guided by Dynamic Indices of Preload Responsiveness Monitoring on Postoperative Complications in Major Hepatic Surgery for Primary or Secondary Liver Cancer
Brief Title: Cardiac Output Optimization on Postoperative Complications in Major Hepatic Surgery
Acronym: OPTILIVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OPTILIVER TRIAL-IPC 2018-022
Record Dates: First submitted 2020-11-27; First posted 2020-12-07 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Primary or Metastatic Hepatic Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimization of cardiac flow by base water-electrolyte supply (Experimental): Optimization of cardiac flow by base water-electrolyte supply of 1 ml / kg / h by Ringer Lactate® and faced with any decrease of more than 10% of the VES compared to the reference VES, achievement of an optimization of the preload by administration of 250 ml of Ringer Lactate® with renewal until correction of the VES.
  Interventions: Behavioral: Optimization of cardiac flow by base water-electrolyte supply
- Control arm (Other): Increase basic hydro-electrolyte supply of 6 ml / kg / h by Ringer Lactate® and 1: 1 blood loss compensation by crystalloids of the same nature.
  Interventions: Behavioral: Control arm

INTERVENTIONS:
Behavioral: Optimization of cardiac flow by base water-electrolyte supply — optimization of cardiac flow by base water-electrolyte supply of 1 ml / kg / h by Ringer Lactate® and faced with any decrease of more than 10% of the VES compared to the reference VES, achievement of an optimization of the preload by administration of 250 ml of Ringer Lactate® with renewal until correction of the VES.
  Arms: Optimization of cardiac flow by base water-electrolyte supply
Behavioral: Control arm — increase basic hydro-electrolyte supply of 6 ml / kg / h by Ringer Lactate® and 1: 1 blood loss compensation by crystalloids of the same nature.
  Arms: Control arm

SUMMARY:
Major hepatectomies are high-risk surgeries offered more and more frequently for the curative treatment of primary or secondary liver cancer, and for complex cases, representing a real challenge for medical teams. The 1st peroperative phase of "hepatic resection" requires a minimum supply of filling fluids to limit perioperative bleeding (Low Central Venous Pressure). However this strategy exposes the risk of organ hypoperfusion due to low cardiac flow, secondary to hypovolaemia, which may lead to ischemic situations favoring the onset of postoperative complications. On the other hand, the hemodynamic management of the 2nd peroperative phase "post hepatic resection" is marked by the need to correct this hypoperfusion by optimizing cardiac output by suitable vascular filling.

The major challenge is thus to restore cardiac output by refilling without excess, by correcting the hypovolemia that arose during the "post resection of the hepatic parenchyma" phase.

Our hypothesis is that an individualized protocol for optimizing intraoperative cardiac flow by guided vascular filling during the "post hepatic resection" phase is accompanied by a reduction in postoperative complications in patients operated on for major hepatic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old,
2. Signature of consent,
3. Any patient scheduled for major hepatic surgery (≥ 3 segments) scheduled by laparotomy, for primary hepatic cancer or secondary metastases,
4. Affiliation to the ''National security'' regimen or beneficiary of this regimen.

Exclusion Criteria:

1. Emergency surgery,
2. Cirrhosis: depending on availability of CT and / or MRI imaging results, clinical examination, Biology (PT, Bilirubin) or histological results (preoperative biopsies in healthy liver)
3. Portal hypertension: depending on availability of imaging data, history of esophageal varices
4. Contraindication to fitting a tool for monitoring dynamic hemodynamic indices (case of esophageal varices for esophageal Doppler for example),
5. Benign tumors,
6. Associated procedures programmed at the same operating time (excluding hepatic surgery): programmed associated digestive resection (colorectal or pancreatic),
7. Laparoscopy,
8. Liver transplantation,
9. Woman pregnant or likely to be (without effective contraception) or breastfeeding,
10. Person in an emergency situation, adult person subject to a legal protection measure (adult under guardianship, guardianship or legal protection), or unable to express consent,
11. Inability to undergo medical monitoring of the trial for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the cardiac output optimization strategy on the occurrence of postoperative complications | From Day 1 to Day 30 post-surgery
  Assessment of the impact of an individualized protocol for optimizing perioperative cardiac flow guided by monitoring of dynamic indices of preload dependence during the post-hepatic resection phase on the occurrence of postoperative complications in major hepatic surgery, for primary hepatic cancer or metastatic origin. We retain as the primary endpoint, the percentage of patients with at least one postoperative complication regardless of the grade in the Dindo-Clavien classification.

SECONDARY OUTCOMES:
Evaluation of grade III-IV postoperative complication in the Dindo-Clavien classification | From Day 1 to Day 30 post-surgery
  To determine whether the strategy for optimizing cardiac output guided by dynamic dependence preload indices is associated with a difference in the incidence of occurrence of at least one grade III-IV postoperative complication in the Dindo-Clavien classification
Evaluation of length of stay in the hospital | From Day 1 to Day 30 post-surgery
  To determine whether the cardiac output optimization strategy guided by the dynamic dependence preload indices is associated with a difference in the length of stay in the Continuing Care Unit, intensive care unit or length of hospital stay or on re-hospitalization rates
Evaluation of mortality | On Day 1, Day 30 and Day 90 post-surgery
  To determine whether the cardiac output optimization strategy guided by the dynamic dependence preload indices is associated with a difference in mortality at D30 and D90
Evaluation occurrence of organ failures | From Day 1 to Day 7 post-surgery
  To determine whether the cardiac output optimization strategy guided by dynamic dependence preload indices has an impact on the occurrence of organ failures, which will be evaluated by the SOFA score per device from Day 1 to Day 7 postoperatively
Evaluation of hemodynamic parameters | From Day 0 to Day 1 post-surgery
  To determine whether the cardiac output optimization strategy guided by dynamic dependence preload indices is associated with a difference on hemodynamic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Manuel de Guibert, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France